CLINICAL TRIAL: NCT04175275
Title: Middle Ear Implant: Assessment of Satisfaction in the Medium Term
Acronym: IOM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0283
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview patient — Interview patient without scoring about the reasons for the implant, the complications, the reasons for abandonment, the evaluation of the satisfaction

SUMMARY:
Currently, the data from the literature do not evaluate the use of the middle ear implant in implanted patients in the medium term (10 years and over) but only in the short term (1-5 years).

Based on the observation of the absence of these data, we considered it necessary to evaluate in the medium term the satisfaction of the patients carrying a middle ear implant and their rate of abandonment with a horizon of 10 to 20 years of apparatus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient accepting to participate to this study
* Patient having a middle ear implant since 10 - 20 years at time of inclusion

Exclusion Criteria:

* patient not dead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all living patients who have benefited from the placement of a middle ear implant since 1998 at Hospices Civils of Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
the abandonment rate | at inclusion
  calculate the rate of patient having abandonment the Use of Middle Ear Implant

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, MD, Principal Investigator — Service de chirurgie ORL et cervico faciale
Locations (1):
- Hopital Edouard Herriot, Lyon, France